CLINICAL TRIAL: NCT06691269
Title: Evaluation of a Photobiomodulation Device for Dental Analgesia in Pediatric Patients
Brief Title: Photobiomodulation and Tooth Analgesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: HP-00112812; Project ID: 30063251 (Other: University of Maryland, Baltimore)
Record Dates: First submitted 2024-10-31; First posted 2024-11-15 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Dental Anaesthesia; Dental Pain; Dental Analgesia
Keywords: photobiomodulation; dental analgesia; dental anesthesia
MeSH Terms: conditions — Toothache | interventions — Low-Level Light Therapy; Benzocaine; Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Study Design: This will be a series of three prospective, clinical studies in school-aged children requiring routine dental procedures.
  Study Population: Healthy children aged 6-12 years old requiring routine dental treatment at the study sites. Separate cohorts will be recruited for each trial after obtaining parental consent.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- PBM- Study 1 (Experimental): In PBM group, the selected tooth will receive one burst of light application (20 seconds) before being subjected to sensibility testing and gingival probing.
  Interventions: Device: Photobiomodulation
- no PBM - Study 1 (No Intervention): In the control (no PBM) group, the selected tooth will be subjected to sensibility testing and gingival probing without PBM.
- PBM- Study 2 (Experimental): PBM (one burst/ 20 seconds application) at injection site (prior to local anesthesia infiltration)
  Interventions: Device: Photobiomodulation
- no PBM- Study 2 (Active Comparator): Topical benzocaine at injection site (prior to local anesthesia infiltration)
  Interventions: Drug: Topical Benzocaine
- PBM- Study 3 (Experimental): PBM (one burst/ 20 seconds application) followed by traditional tooth preparation with burs/handpiece and placement of restoration. Additional bursts may be provided every 20 minutes depending on the length of the procedure and patient-reported discomfort.
  Interventions: Device: Photobiomodulation
- no PBM- Study 3 (Active Comparator): Topical benzocaine/Local infiltration followed by traditional tooth preparation with burs/handpiece and placement of restoration.
  Interventions: Drug: Topical Benzocaine; Drug: Local Anesthesia

INTERVENTIONS:
Device: Photobiomodulation — Photomodulation (PBM) is a promising non-tissue penetrating (i.e. minimally invasive) approach for achieving tooth and soft tissue anesthesia/analgesia in dental patients. A patent pending near-infrared laser technology that aims to provide dental analgesia will be used for PBM. This intra-oral PBM device comes with a tip comprising of a series of photonic emitters with specific wavelengths that can go through the tooth structure and bone, blocking the nerve conduction like local anesthetics. Research has shown that one burst of light application (for about 20 second) can provide up to 15-20 minutes of pain relief. Based on existing research PBM does not present a serious risk to health, safety, or welfare of a subject.
  Other Names: Low-level light therapy, near-infrared light
  Arms: PBM- Study 1; PBM- Study 2; PBM- Study 3
Drug: Topical Benzocaine — Topical Benzocaine at injection site to reduce discomfort of local infiltration
  Arms: no PBM- Study 2; no PBM- Study 3
Drug: Local Anesthesia — Local infiltration using local anesthetics with epinephrine
  Arms: no PBM- Study 3

SUMMARY:
The purpose of this study is to test photobiomodulation (PBM) with a non-invasive light device for reducing discomfort during dental treatments in children. We plan to conduct a series of three clinical studies in 200 school-aged children requiring routine dental treatment. The first study aims to test if PBM works for tooth and soft tissue by assessing response to cold testing and probing of gums. The second study aims to test if use of PBM on soft tissues before injection reduces discomfort. The third study aims to test if PBM can be used to do simple dental fillings in baby teeth without numbing injection.

DETAILED DESCRIPTION:
Dental anxiety and fear of pain during procedures are major barriers to oral health care, especially among children. Traditional local anesthesia injections can be distressing for pediatric patients. The fear of needle and dental pain are perhaps among the top reasons for avoidance of dental care. Photomodulation (PBM) is a promising non-tissue penetrating (i.e. minimally invasive) approach for achieving tooth and soft tissue anesthesia/analgesia in dental patients.Investigators plan to use an intra-oral PBM device with a tip comprising of a series of photonic emitters with specific wavelengths that can go through the tooth structure and bone, blocking the nerve conduction like local anesthetics. Research has shown that one burst of light application (for about 20 second) can provide up to 15-20 minutes of pain relief. This could significantly reduce dental anxiety and facilitate access to care and the implications of such an alternative to needles will be a gamechanger especially in pediatric dentistry. The proposed randomzied clinical trials will evaluate if photobiomodulation (PBM) with the near-infrared device produces dental analgesia comparable to local anesthetic injection in pediatric patients. This will be a series of three prospective, clinical studies in 200 school-aged children aged 6-12 years requiring routine dental procedures. The first trial will test the effectiveness of PBM in tooth and soft tissue analgesia by assessing response to diagnostic approaches such as cold pulp testing and gingival probing. The second trial will assess the pre-emptive analgesic effect of PBM on soft tissues at the site of injection prior to local anesthesia infiltration to reduce the discomfort of injection, and the third trial will assess effectiveness of PBM in providing tooth analgesia (compared to routinely used topical anesthesia/local infiltration) for simple restorative procedures in primary teeth.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children, aged 6-12 years, requiring routine dental treatment

Exclusion Criteria:

* Children with uncooperative behavior or signficant medical history

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Study 1- Response to Cold Pulp (Pulp sensibility) testing | during the intervention (application of cold stimuli)
  Name of measurement: Response to cold pulp testing. Measurement tool: Child's acknowledgement of cold sensation. A small amount of cold spray (Endo Ice/Ethyl Chloride) will be sprayed onto a cotton pellet, and gently place the cotton pellet on the middle third of the buccal surface of the tooth for a few seconds or until the child indicates a sensation. Child will be asked to raise their hand when they feel a cold sensation.
  Unit of measurement: Response will be noted (Yes/No), if the cold sensation is felt by the child on application of cold stimulus. Difference in cold pulp testing between PBM and no PBM group.
Study 1- Anxiety related to routine gingival probing | pre-procedure (baseline) and immediately after the procedure
  Name of the measurement: Assessment of anxiety Measurement tool: Visual analogue scale (VAS)- a 100-mm horizontal line with two extremes "not anxious" (left) to "very anxious" (right).
  Measurement unit: rating scale
Study 1- Pain (physician documented) related to routine gingival probing | pre-procedure (baseline), during procedure, and immediately after procedure
  Name of the measurement: Heart rate Measurement tool: Pulse oximetry. Unit of measurement: Heart rate per minute
Study 1- Self-reported Pain related to routine gingival probing | pre-procedure (baseline) and immediately after procedure
  Name of the measurement: Pain/discomfort Measurement tool: Self-reported Wong Baker faces Scale (six-point scale from score 0 (no hurt) to score 10 (hurts worst).
  Unit of measurement: Rating Scale
Study 2- Anxiety related to local anesthesia injection (local infiltration) | pre-procedure (baseline) and immediately after the procedure
  Name of the measurement: Assessment of procedural anxiety Measurement tool: Visual analogue scale (VAS)- a 100-mm horizontal line with two extremes "not anxious" (left) to "very anxious" (right).
  Measurement unit: rating scale
Study 2- Pain (physician documented) related to local anesthesia injection (local infiltration) | pre-procedure (baseline), during procedure, and immediately after procedure
  Name of the measurement: Heart rate Measurement tool: Pulse oximetry. Unit of measurement: Heart rate per minute
Study 2- Self-reported Pain related to local anesthesia injection (local infiltration) | pre-procedure (baseline) and immediately after procedure
  Name of the measurement: Pain/discomfort Measurement tool: Self-reported Wong Baker faces Scale (six-point scale from score 0 (no hurt) to score 10 (hurts worst).
  Unit of measurement: Rating Scale
Study 2- Cooperative behavior related to local anesthesia injection (local infiltration) | pre-procedure (baseline), during, and immediately after procedure
  Name of the measurement: Cooperative behavior Measurement tool: Frankel's Behavior rating scale (definitely negative, negative, positive, definitely positive) Unit of measurement: Rating Scale
Study 3- Anxiety during restorative procedure | pre-procedure (baseline) and immediately after the procedure
  Name of the measurement: Assessment of procedural anxiety Measurement tool: Visual analogue scale (VAS)- a 100-mm horizontal line with two extremes "not anxious" (left) to "very anxious" (right).
  Measurement unit: rating scale
Study 3- Pain (physician documented) during restorative procedure | pre-procedure (baseline), during procedure, and immediately after procedure
  Name of the measurement: Heart rate Measurement tool: Pulse oximetry. Unit of measurement: Heart rate per minute
Study 3- Self-reported Pain during restorative procedure | pre-procedure (baseline) and immediately after procedure
  Name of the measurement: Pain/discomfort Measurement tool: Self-reported Wong Baker faces Scale (six-point scale from score 0 (no hurt) to score 10 (hurts worst).
  Unit of measurement: Rating Scale
Study 3- Cooperative behavior during restorative procedure | pre-procedure (baseline), during, and immediately after procedure
  Name of the measurement: Cooperative behavior Measurement tool: Frankel's Behavior rating scale (definitely negative, negative, positive, definitely positive) Unit of measurement: Rating Scale

SECONDARY OUTCOMES:
Study 1- Duration of tooth analgesia in PBM group | baseline and immediately after response is felt
  Name of measurement: Duration or time taken for response to cold pulp testing. Measurement tool: Child's acknowledgement of cold sensation. A small amount of cold spray (Endo Ice/Ethyl Chloride) will be sprayed onto a cotton pellet, and gently place the cotton pellet on the middle third of the buccal surface of the tooth for a few seconds or until the child indicates a sensation. Child will be asked to raise their hand when they feel a cold sensation.
  Unit of measurement: Time (measured in seconds) taken for response in PBM group and no PBM groups.
Study 1- Duration of soft tissue analgesia | baseline, immediately after response is felt
  Name of measurement: Duration of analgesia or time taken for patient to respond to gingival probing Measurement tool: Yes/No to discomfort experienced during gingival probing Unit of measurement: Time in seconds

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Dentistry, Pediatric Clinics, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shrutha SP, Havale R, Aishwarya BG, Raj S, Quazi N, Prasad V, Guttiganur N, Kandalam R. Use of Three Pre-Injection Procedures to Reduce Pain Perception of Intraoral Injections in Eight- to 12-Year-Old Children: Randomized Controlled Trial. Pediatr Dent. 2024 Sep 15;46(5):306-311. PMID 39420491
- [Result] Shekarchi F, Nokhbatolfoghahaei H, Chiniforush N, Mohaghegh S, Haeri Boroojeni HS, Amini S, Biria M. Evaluating the Preemptive Analgesic Effect of Photo-biomodulation Therapy on Pain Perception During Local Anesthesia Injection in Children: A Split-mouth Triple-blind Randomized Controlled Clinical Trial. Photochem Photobiol. 2022 Sep;98(5):1195-1200. doi: 10.1111/php.13605. Epub 2022 Feb 17. PMID 35122442
- [Result] Kulkarni S, George R, Love R, Ranjitkar S. Effectiveness of photobiomodulation in reducing pain and producing dental analgesia: a systematic review. Lasers Med Sci. 2022 Sep;37(7):3011-3019. doi: 10.1007/s10103-022-03590-4. Epub 2022 Jun 14. PMID 35699807